CLINICAL TRIAL: NCT05580159
Title: A Multi-national, Randomized, Observer-blinded, Parallel Controlled Trial to Evaluate the Immunogenicity and Safety of New Generation COVID-19 mRNA Booster Vaccination Against Emerging Variants of Concern (VOC)
Brief Title: New Generation mRNA Booster Vaccine Against Emerging VOCs
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stemirna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SWC310
Record Dates: First submitted 2022-10-08; First posted 2022-10-14 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Immunogenicity; Efficacy; Safety
Keywords: new generation mRNA vaccine

STUDY DESIGN:
Intervention Model Description: a randomized observer-blinded parallel controlled trial：Experimental group（mRNA vaccine） and positive control group（inactive vaccine）
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study uses a double blinded design, and the investigators and participants will all remain blinded before unblinding and do not know which group the participant belongs to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SW-BIC-213 (Experimental): Intervention Name :COVID-19 mRNA vaccine Type :Investigational Vaccine Dose :Formulation mRNA Unit Dose Strength(s) :0.5ml; Dosage Level(s) :0.25ml; Route of Administration: injection Intramuscular
  Interventions: Biological: SW-BIC-213
- SARS-Cov-2 Vaccina(Vero Cell ) Inactivated (Active Comparator): Intervention Name: COVID-19 Inactivated Vaccine Type : Control Vaccine Dose :Inactive Unit Dose Strength(s) : 0.5ml; Route of Administration Intramuscular : injection Intramuscular
  Interventions: Biological: SARS-Cov-2 Vaccina(Vero Cell ) Inactivated

INTERVENTIONS:
Biological: SW-BIC-213 — The patient will take a single 25 μg dose mRNA vaccine SW-BIC-213.
  Arms: SW-BIC-213
Biological: SARS-Cov-2 Vaccina(Vero Cell ) Inactivated — The patient will take a third dose of COVID-19 Inactivated vaccine.
  Arms: SARS-Cov-2 Vaccina(Vero Cell ) Inactivated

SUMMARY:
Primary：Objectives ：SafetyTo describe the safetyprofile of all participants in each group up to 6months post-dose.Immunogenicity：To demonstrate the superiorityof neutralizing antibodyresponse in terms of geometric mean titers (GMT) of mRNA vaccine compare with inactive vaccine28 days post dose. Secondary:Immunogenicity

1. To describe binding antibodyprofile at D01,D08, D15, D29,D91 and D181 of eachstudy group.
2. To describe the neutralizing antibody profile atD08,D15,D91 and D181of 600 participants for each studyintervention group. Exploratory:Cell-mediated immunity To describe the cellular immuneresponse profile at D01, D08, D15and D29, in a subset of 30 participants for each study group.

Efficacy:To describe the occurrence of virologically-confirmed COVID-19 like illness and serologically confirmed SARS-CoV-2 infection.

DETAILED DESCRIPTION:
Endpoints:Safety Endpoints- Occurrence of unsolicited systemic AEs reported in the 30 minutes after each injection.

Occurrence of solicited injection site reactions and systemicreactions occurring up to 7 days post-dose.

Occurrence of unsolicited non-serious AEs reported up to 28 dayspost-dose. Occurrence of SAEs and AESIs up to 6 months throughout the study. Immunogenicity Endpoints:GMT of neutralizing antibody will be measured with the neutralization assayon D01,D29.

Binding antibody titers to full length SARS-CoV-2 Spike (S) protein will be measured for each study intervention group with the ELISA method

* Antibody titer on D01, D08, D15, D29, D91, D181
* Fold-rise in antibody titer at D08, D15, D29, D91 and D181 post vaccination relative to D01
* 4-fold-rise in antibody titer at D08, D15, D29, D91, and D181 relative to D01 Neutralizing antibody titers will be measured with the neutralization assay
* Antibody titer on D08, D15, D29, D91 and D181
* Fold-rise (fold rise in serum neutralization titer post vaccination relative to D01) at D08, D15, D29, D91 and D181
* 4-fold rise in serum neutralization titer [post/pre] relative to D01 at D08, D15, D29, D91 and D181
* Occurrence of neutralizing antibody seroconversion, defined as baseline values below LLOQ at baseline with detectable neutralization titer above assay lower limit of quantification at D08, D15, D29, D91 and D181INF-γ, IL-4 and IL-2 will be measured in whole blood and/or cryopreserved PBMC following stimulation with pools of S
* ExploratoryCell-mediated immunity To describe the cellular immune response profile at D01, D08, D15 and D29, in a subset of 30 participants for each study group antigen peptides.

Virologically-confirmed COVID 19 like illness as defined by specified clinical symptoms and signs and confirmed by a positive result for SARS-CoV-2 nucleic acid viral detection assay.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give written informed consent for participation in the study.
2. Male or Female, aged 18 years or above and in good health as determined by study clinician.
3. Female participants of childbearing potential must be willing to ensure that they or their partner use effective contraception from 1 month prior to first immunization continuously until 3 months after boost immunization.
4. In the Investigator's opinion, is able and willing to comply with all trial requirements.
5. Subjects had completed the 2-dose series vaccination of COVID-19 inactivated vaccine at least .

24 weeks with the completed the 2-dose Series as the primary vaccination according to the product label.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

1. Confirmed cases, suspected cases or asymptomatic cases of COVID-19;
2. Self-reported history of SARS and MERS infection;
3. Receipt of live attenuated vaccine within one month prior to vaccination and other vaccines within 14 days prior to vaccination;
4. Receipt of any SARS-COV-2 vaccine after last dose of primary vaccination
5. Participants who are pregnant at enrolment or planning to become pregnant during the first 3 months following vaccination.
6. Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccines.
7. History of allergic disease or reactions likely to be exacerbated by any component of study vaccines.
8. Any history of anaphylaxis to any component of vaccine.
9. Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or continuous use of anticoagulants (warfarin, apixaban, rivaroxaban, dabigatran, edoxaban), or prior history of significant bleeding or bruising following IM injections or venipuncture.
10. Suspected or known current alcohol or drug dependency
11. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
12. Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, and neurological illness (mild/moderate well controlled comorbidities are allowed).
13. Scheduled elective surgery during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-05-11 (Estimated); Study Completion 2023-05-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 6 months post-dose
  To describe the safety profile of all participants in each group up to 6 months post-dose.
Immunogenicity of 28 days post dose | 28 days post dose
  To demonstrate the superiority of neutralizing antibody response in terms of geometric mean titers (GMT) of mRNA vaccine compare with inactive vaccine 28 days post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Mayfong Mayxay, doctor, Principal Investigator — National Ethics Committee for Health Research(NECHR)
Locations (1):
- Savannakhét Provincial hospital, Savannakhet, Sava, Laos

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fang Y, Li JX, Duangdany D, Li Y, Guo XL, Phamisith C, Yu B, Shen MY, Luo B, Wang YZ, Liu SJ, Zhao FF, Xu CC, Qiu XH, Yan R, Gui YZ, Pei RJ, Wang J, Shen H, Guan WX, Li HW, Mayxay M. Safety, immunogenicity, and efficacy of a modified COVID-19 mRNA vaccine, SW-BIC-213, in healthy people aged 18 years and above: a phase 3 double-blinded, randomized, parallel controlled clinical trial in Lao PDR (Laos). EClinicalMedicine. 2023 Dec 13;67:102372. doi: 10.1016/j.eclinm.2023.102372. eCollection 2024 Jan. PMID 38169790